CLINICAL TRIAL: NCT02925624
Title: 'CLOSE'-Guided Pulmonary Vein Isolation as Cure for Paroxysmal Atrial Fibrillation?
Brief Title: CLOSE to CURE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Prof. Dr. Mattias Duytschaever, Professor Doctor, AZ Sint-Jan AV
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1949
Record Dates: First submitted 2016-09-29; First posted 2016-10-06 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation
Keywords: ablation index; pulmonary vein isolation; implantable loop recorder
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CLOSE guided PVI and insertable cardiac monitor (Experimental)
  Interventions: Procedure: Pulmonary vein isolation

INTERVENTIONS:
Procedure: Pulmonary vein isolation

SUMMARY:
Title: CLOSE-guided pulmonary vein isolation (PVI) as Cure for Paroxysmal Atrial Fibrillation ('CLOSE to CURE' study)

Design: This is a prospective, observational, single-center, unblinded, clinical 3-year study.

Background: In a population of paroxysmal atrial fibrillation (AF) 'CLOSE'-guided PVI, a new approach to obtain single-procedure durable PVI, has been shown to virtually eliminate recurrence of AF at 1 year follow-up with repetitive but discontinuous Holter monitoring.

Objectives: (1) To objectively compare atrial tachyarrhythmia (ATA) burden before and after 'CLOSE'-guided based PVI using continuous monitoring. (2) To assess ATA burden using continuous monitoring up to 3 years after ablation. (3) To identify baseline structural and electrical properties of the atria or procedural characteristics that predict 1-year and 3-year outcome.

Enrollment: Up to 100 subjects will be enrolled in this observational, prospective study.

Clinical Sites: 1 site.

Subject Population: Eligible patients are patients with paroxysmal high-burden AF who are planned for a 'CLOSE'-guided PV isolation. At the time of procedural planning we will ask the patient his/her consent for (1) implantation of a subcutaneous continuous loop recorder (sCLR), (2) a concise electrophysiological study at the time of PVI, (3) a transthoracic echocardiogram at the time of PVI and (4) collection of data during 3 years. Anti-arrhythmic drug treatment (ADT) and oral anticoagulation (OAC) will be given according the updated 2012 European society of Cardiology (ESC) guidelines on AF (Camm et al, European Heart Journal 2012) and the 2012 Heart rhythm society (HRS)/European Heart Rhythm association/European cardiac arrhythmic society Expert Consensus Statement on catheter and surgical ablation of atrial fibrillation (Calkins et al, Heart Rhythm 2012).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic paroxysmal AF (history of self-terminating AF within 7 days or history of self-terminating AF with 1 or more cardioversions within 48 hours after onset), meeting following criteria at the out-patient clinic:

   * patient has at least 3 AF episodes in the last 3 months prior to the visit
   * AF episodes are symptomatic, and patient is drug-resistant (at least one class IC or III), or drug-intolerant (palpitations, fatigue, dyspnea, cardiomyopathy,…)
   * no advanced structural heart disease
   * patient has a CHA2DS2-VASc score of 0, 1, 2, 3 or 4
2. Signed Patient Informed Consent Form.
3. Age 18 years or older.
4. Able and willing to comply with all follow-up testing and requirements.

Exclusion Criteria:

1. Persistent atrial fibrillation (history of AF>7days or history of cardioversion > 48h of AF)
2. Previous ablation for AF
3. LA antero-posterior diameter > 50 mm (parasternal long axis view , PLAX)
4. LVEF < 35% (ejection fraction)
5. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
6. Coronary artery bypass grafting (CABG) procedure within the last three months
7. Awaiting cardiac transplantation or other cardiac surgery
8. Documented left atrial thrombus on imaging
9. Diagnosed atrial myxoma
10. Women who are pregnant or breastfeeding
11. Acute illness or active systemic infection or sepsis
12. Unstable angina
13. Uncontrolled heart failure
14. Myocardial infarction within the previous two months
15. History of blood clotting or bleeding abnormalities
16. Contraindication to anticoagulation therapy (ie, heparin or warfarin)
17. Life expectancy less than 12 months
18. Enrollment in any other study evaluating another device or drug
19. Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-12; Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Atrial tachyarrhythmia (ATA) burden before and after 'CLOSE'-guided based PVI | Continuous monitoring (24 hours loop recording)
Long-term evaluation of ATA burden after a single 'CLOSE' guided PVI procedure | Continuous monitoring (24 hours loop recording)

SECONDARY OUTCOMES:
Evaluating PV re-connection at redo procedure assessed by Lasso catheter | 3 months to 3 years
  Visual inspection of electrograms on the Lasso catheter will be performed to verify durable PV isolation or re-connection
Evaluating progression of scarring at redo procedure assessed by voltage mapping | 3 months to 3 years
  Point-by-point bipolar voltage mapping will be performed to quantify the amount of low voltage areas in the left atrium (LA)
Incidence of adverse events related to ablation | Baseline to 3 years
Freedom from stroke/transient ischemic attack (TIA) | Baseline to 3 years
Efficacy of CLOSE protocol ablation assessed by single-procedure freedom from documented atrial tachyarrhythmias (ATA) | 1 month to 3 years
  ATA include fibrillation, tachycardia, or flutter
Efficacy of CLOSE protocol ablation assessed by incidence of repeat ablation procedures | 1 month to 3 years
Efficacy of CLOSE protocol ablation assessed by multiple-procedure freedom from ATA | 1 month to 3 years
  ATA include fibrillation, tachycardia, or flutter
Health economics and outcomes research assessed by quality of life using Short Form (SF-36v2) Health Survey | Recruitment to 3 years
Health economics and outcomes research assessed by quality of life using Symptomatic Questionnaire V3 | Recruitment to 3 years
Health economics and outcomes research assessed by number of hospitalization | Recruitment to 3 years
  Includes total number of hospitalizations and unscheduled arrhythmia-related health care provider visits

OTHER OUTCOMES:
Clinical characteristic assessed by height | At baseline
Clinical characteristic assessed by weight | At baseline
Clinical characteristic assessed by age | At baseline
Clinical characteristic assessed by sex | At baseline
Clinical characteristic assessed by congestive heart failure history | At baseline
Clinical characteristic assessed by hypertension history | At baseline
Clinical characteristic assessed by stroke/TIA/Thromboembolism history | At baseline
Clinical characteristic assessed by vascular disease history | At baseline
Clinical characteristic assessed by diabetes mellitus | At baseline
Clinical characteristic assessed by left ventricle ejection fraction (LVEF) | At baseline
Clinical characteristic assessed by structural heart disease | At baseline
Clinical characteristic assessed by endurance measured by amount of training/cycling per week | At baseline
Clinical characteristic assessed by history of implanted devices | At baseline
Clinical characteristic assessed by LA diameter measured by echocardiography | At baseline
Clinical characteristic assessed by LA volume measured by echocardiography | At baseline
Clinical characteristic assessed by cardiovascular medication history | At baseline
Procedure characteristic assessed by procedure time | At baseline
Procedure characteristic assessed by radiofrequency time | At baseline
Procedure characteristic assessed by fluoroscopy time | At baseline
Electrophysiological characteristic assessed by voltage mapping of the LA | At baseline
  Point-by-point bipolar voltage mapping will be performed to quantify the amount of low voltage areas in the LA
Electrophysiological characteristic assessed by atrial refractoriness | At baseline
  This will be done by premature stimulation protocol
Electrophysiological characteristic assessed by conduction velocity | At baseline
  This will be done by premature stimulation protocol
Electrophysiological characteristic assessed by AF inducibility | At baseline
  This will be done by premature stimulation protocol

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Duytschaever, MD, PhD, Principal Investigator — Department of Cardiology, AZ Sint-Jan Hospital Bruges, Belgium
Locations (1):
- AZ Sint-Jan Hospital, Bruges, Belgium

REFERENCES:
- [Derived] Duytschaever M, De Pooter J, Demolder A, El Haddad M, Phlips T, Strisciuglio T, Debonnaire P, Wolf M, Vandekerckhove Y, Knecht S, Tavernier R. Long-term impact of catheter ablation on arrhythmia burden in low-risk patients with paroxysmal atrial fibrillation: The CLOSE to CURE study. Heart Rhythm. 2020 Apr;17(4):535-543. doi: 10.1016/j.hrthm.2019.11.004. Epub 2019 Nov 9. PMID 31707159